CLINICAL TRIAL: NCT00163735
Title: Potential Allergens in Wine: Double Blind Placebo-controlled Trial and Basophil Activation Analysis
Brief Title: Potential Allergens in Wine: Double-blind Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Australian Wine Research Institute (Other); National Health and Medical Research Council, Australia (Other); The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 124/02; Number 124/02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Food Allergy; Anaphylaxis
Keywords: Food allergy; wine; milk allergy; egg allergy; nut allergy; fish allergy
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis; Milk Hypersensitivity; Egg Hypersensitivity; Nut Hypersensitivity

INTERVENTIONS:
Drug: Administration of wine fined with potential food allergens

SUMMARY:
This study is designed to identify whether wines which are produced using the common potential food allergens such as proteins derived from fish, milk or egg are likely to contain sufficient food allergens to cause allergic reactions in susceptible individuals.

DETAILED DESCRIPTION:
Recent international legislation requires labelling of wines made using potentially allergenic food proteins "casein", egg white, isinglass ( fish derived), milk or evaporated milk where "there is detectable residual processing aid". However it is not clear whether the final wine contains concentrations of residual added food proteins that can provoke allergic reactions.

Comparison:This study is a double blind, placebo-controlled trial to determine whether adults known to be allergic to eggs, fish, milk and/or nuts exhibit allergic reactions following consumption of Australian commercial wines fined with food allergens.

ELIGIBILITY:
Inclusion Criteria:

Individuals with IgE-mediated food allergy to milk, fish, egg or nuts Otherwise no major medical problems Able to drink wine -

Exclusion Criteria:

Major asthma or cardiac disease Unwilling or unable to participate

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Allergic reactions to wine

SECONDARY OUTCOMES:
Positive basophil activiation test to wines

CONTACTS AND LOCATIONS:
Overall Officials: Robyn E O'Hehir, MBBS PhD FRACP, Study Director — Alfred Hospital and Monash University; Jennifer M Rolland, PhD, Principal Investigator — Monash University; Creina S Stockley, PhD, Principal Investigator — The Australian Wine Research Institute
Locations (1):
- AIR Med, Alfred Hospital, Melbourne, Victoria, Australia